CLINICAL TRIAL: NCT02182596
Title: A Dose-finding Phase I/II Trial of Daunorubicin and Cytarabine Combined to Fractionated Mylotarg® as Re-induction Treatment in Patients With First Relapse of Acute Myeloid Leukemia
Brief Title: DNR and AraC Combined to Fractionated Mylotarg® in Patients With First Relapse of AML
Acronym: MYLOFRANCE2
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Acute Leukemia French Association (Other)
Responsible Party: Pr Sylvie CASTAIGNE, VERSAILLES HOSPITAL
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MYLOFRANCE 2
Record Dates: First submitted 2011-01-19; First posted 2014-07-08 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute Myeloid Leukemia; First relapsing AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Gemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- DAUNORUBICINE - ARACYTINE - MYLOTARG - (Experimental): Adaptive Bayesian method for dose-finding in phase I/II clinical trials based on treatment efficacy and toxicity (Thall, Russel, 1998), with successive patients cohorts and three combined dose levels:
  DNR 45 mg/m2 IV days 1 to 3 + AraC 100 mg/m2 CI days 1 to 7 + Mylotarg 3mg/m2 IV days 1, 4, 7.
  DNR 60 mg/m2 IV days 1 to 3 + AraC 100 mg/m2 CI days 1 to 7 + Mylotarg 3mg/m2 IV days 1, 4, 7.
  DNR 60 mg/m2 IV days 1 to 3 + AraC 200 mg/m2 CI days 1 to 7 + Mylotarg 3mg/m2 IV days 1, 4, 7.
  Two consolidation courses for CR patients:
  Amsacrine: 90 mg/m2 IV Day 1 Cytarabine: 1g/m2 twice a day IV Days 1 to 4 Mylotarg: 3 mg/m2 IV Day 1.
  Interventions: Drug: Mylotarg

INTERVENTIONS:
Drug: Mylotarg — Dose level study
  Other Names: Gemtuzumab Ozogamicin

SUMMARY:
For several years, the effective standard induction chemotherapy for AML has been limited to the association of anthracycline and aracytine. GO is the first effective targeted antibody used in leukemia patients. In a previous study, we showed efficacy and safety of fractionated doses of GO used as a single agent for treatment of adult AML patients in first relapse. In the present study the possibility of combining fractionated doses of GO to escalated doses of a 3+7 regimen old is studied in relapsed AML patients > 50 and <70 years.

DETAILED DESCRIPTION:
Induction course are:

GO 3mg/m2 on days 1, 4,7 + the three dose levels were as follows:

level 1: DNR: 45 mg/m2 x 3 days + AraC: 100 mg/m2 x 7 days level 2: DNR: 60 mg/m2 x 3 days + AraC: 100 mg/m2 x 7 days level 3: DNR 60 mg/m2 x 3 days + AraC: 200 mg/m2 x 7 days. with 20 mg of methylprednisolone prior to each GO infusion. Consolidation course: patients in CR may receive 2 additional courses of consolidation chemotherapy with Amsacrine 90 mg/m2 daily for 3 days, and Ara-C (1g/m2/12 hours x 3 days) + GO 3 mg/m2 on day 1.

Treatment with HSCT is offered at the discretion of the physician in charge of the patient. A delay between last infusion of GO and HSCT above 3 months is recommended

ELIGIBILITY:
Inclusion Criteria:

Patients with a morphologically proven diagnosis of CD33-positive AML and :

1. Age ≥ 50 years and ≤ 70 years.
2. First relapsing AML with a duration of first CR ≥ 3 and ≤18 months
3. ECOG performance status 0 to 3
4. Negative serology HIV, HBV and HBC (except post vaccination)
5. Serum creatinine ≤ 2N; AST and ALT ≤ 2N; total bilirubin ≤ 2N
6. Cardiac function determined by radionuclide or echography within normal limits.
7. Negative serum pregnancy test within one week before treatment for women of child bearing potential
8. Signed informed consent.

Exclusion Criteria:

1. M3-AML
2. AML following diagnosed myelodysplastic syndrome or myeloproliferation
3. Known central nervous system involvement with AML
4. Prior treatment with HSCT.
5. Previous treatment with Anti CD33 antibodies
6. Uncontrolled infection
7. Other active malignancy

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-06; Primary Completion 2007-09 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) defined by the occurrence of any G3 or G4 non reversible toxicity at day 45 excluding myelosuppression or infection due to neutropenia, and response defined by complete remission at day 45 | Day 45 post first dose of treatment

SECONDARY OUTCOMES:
Secondary endpoint: Duration of second remission in AML patients treated for relapse with chemotherapy + Mylotarg as re-induction and consolidation. | At two years

CONTACTS AND LOCATIONS:
Overall Officials: CASTAIGNE SYLVIE, PROFESSOR, Principal Investigator — Acute Leukemia French Association
Locations (15):
- France (15):
  - Hopital Avicenne, Bobigny
  - CH, Caen
  - Hopital Percy, Clamart
  - CHU, Créteil
  - CHU, Lille
  - CH, Limoges
  - Hopital Edouard Herriot, Lyon
  - CH, Meaux
  - St Antoine Hospital, Paris
  - Hopital Saint-Louis, Paris
  - CH, Roubaix
  - CHU, Rouen
  - CNLCC, Saint-Cloud
  - CH, Versailles
  - IGR, Villejuif